CLINICAL TRIAL: NCT05177263
Title: Effect of the Different Concentrations of Oral Dextrose Solution Applying Together With Supportive Positions on Pain During the Heel-Stick Sampling in Premature Infants: A Randomized Controlled Study
Brief Title: Effects of the Different Concentrations of Oral Dextrose Solution Applying With Supportive Positions on Pain During Heel-Stick Sampling in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guzide UGUCU (Other)
Responsible Party: Sponsor-Investigator, Guzide UGUCU, Res. Asst., RN, MScN, PhD Candidate, Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MersinU*GUGUCU_002
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Gurmarin protein, Gymnema sylvestre

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The opaque envelopes are stored in a locked cabinet by the researcher who performed the randomization. The group including the eligible premature infants will not be shared care provider and assessors. Parents will be masked to the groups. Data entries will be performed using the codes A, B, C, and D. Codes will be shared with the researchers after statistical analyses are conducted and the research report is written.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Supportive Positions + Oral Sterile Water (Placebo Comparator): The enrolled premature infants will be administered 1ml of the sterile water a first time 2 minutes before the procedure. After 2 minutes, heel-stick sampling (with an auto lancet for premature infants) will be performed immediately after administering 1 ml of sterile water a second time.
  Interventions: Other: Placebo
- Supportive Positions + 10% Oral Dextrose (Active Comparator): The enrolled premature infants will be administered 1ml of the 10% oral dextrose solution a first time 2 minutes before the procedure. After 2 minutes, heel-stick sampling (with an auto lancet for premature infants) will be performed immediately after administering 1 ml of 10% oral dextrose solution a second time.
  (%10 oral dextrose solution: osmolarity= 550 mOsm/L, pH= 3.5-6.5, calorie=400 kcal/L)
  Interventions: Drug: 10% Oral Dextrose Solution
- Supportive Positions + 20% Oral Dextrose (Active Comparator): The enrolled premature infants will be administered 1ml of the 20% oral dextrose solution a first time 2 minutes before the procedure. After 2 minutes, heel-stick sampling (with an auto lancet for premature infants) will be performed immediately after administering 1 ml of 20% oral dextrose solution a second time.
  (%20 oral dextrose solution: osmolarity= 1010 mOsm/L, pH= 3.2-6.5, calorie= 680 kcal/L)
  Interventions: Drug: 20% Oral Dextrose Solution
- Supportive Positions + 30% Oral Dextrose (Active Comparator): The enrolled premature infants will be administered 1ml of the 30% oral dextrose solution a first time 2 minutes before the procedure. After 2 minutes, heel-stick sampling (with an auto lancet for premature infants) will be performed immediately after administering 1 ml of 30% oral dextrose solution a second time.
  (%30 oral dextrose solution: osmolarity= 1515 mOsm/L, pH= 3.2-6.5, calorie= 1020 kcal/L)
  Interventions: Drug: 30% Oral Dextrose Solution

INTERVENTIONS:
Other: Placebo — Sterile Water
  Arms: Supportive Positions + Oral Sterile Water
Drug: 10% Oral Dextrose Solution — 10% Oral Dextrose Solution
  Other Names: Sweet taste
  Arms: Supportive Positions + 10% Oral Dextrose
Drug: 20% Oral Dextrose Solution — 20% Oral Dextrose Solution
  Other Names: Sweet taste
  Arms: Supportive Positions + 20% Oral Dextrose
Drug: 30% Oral Dextrose Solution — 30% Oral Dextrose Solution
  Other Names: Sweet taste
  Arms: Supportive Positions + 30% Oral Dextrose

SUMMARY:
Within the scope of the newborn screening (metabolic and endocrine diseases) tests (NSTs), this research aims to determine the effect of the different concentrations of oral dextrose solution applying together with supportive positions primarily on the pain scores and secondarily on the duration of crying time during the heel-stick sampling in premature infants.

DETAILED DESCRIPTION:
Background Premature infants admitted to the neonatal intensive care unit (NICU) experience pain most frequently due to heel-stick sampling, venipuncture, and peripheral IV placement. The heel-stick method for drawing capillary blood is the most common way to draw newborns' blood. It is used to collect blood for newborn screening tests, usually on the 2nd-7th days after birth. Heel-stick sampling is known to cause moderate to severe pain in premature infants. There is a lack of high-quality evidence in the relevant studies determining effective interventions in the management of pain caused by heel-stick sampling in premature babies.

Research Hypotheses H01: There is no difference in the mean N-PASS scores during the procedure between the groups.

H02: There is no difference in the mean N-PASS scores after the procedure between the groups.

H03: There is no difference in the mean durations of crying after the procedure between the groups.

Design and Settings:This parallel-group randomized trial will be conducted in a Level 4a NICU at a university hospital. For this experimental research, 128 premature infants who will be screened with the routine NSTs are enrolled and randomized into four groups one control group with "supportive positions + oral sterile water (n=32)", one group with "supportive positions + 10% oral dextrose (n=32)", "supportive positions + 20% oral dextrose (n=32)", "supportive positions + 30% oral dextrose (n=32)". The hospital provides education in the field of neonatal nursing (certification) and neonatology (sub-specialty) as a training hospital. The 25-bed unit is one of the tertiary care referral centers in the East Mediterranean Region of Turkey. The admission rate is nearly 214 infants per year on average. Generally, infants come from peripheral (40%), and central (40%) districts, or another city (20%). The unit design is a traditional open-bay type. Heel-stick sampling in premature infants is carried out on the 2nd-10th days after birth within the scope of the NSTs. The Turkish version of the Neonatal Pain Agitation and Sedation Scale (N-PASS) is used as a pain assessment tool in nursing forms. Pain scores of premature infants are evaluated and recorded at each shift change and interventional procedure.

Sample Size: A priori power analysis was used to estimate the sample size based on data from "Brovedani, P., Montico, M., Shardlow, A., Strajn, T., & Demarini, S. (2007). Suckling and sugar for pain reduction in babies. The Lancet, 369(9571), 1429-1430." A priori power analysis was performed based on the effect size (d = 0.929, large effect) of the difference in pain scores between the groups (during the procedure) determined in this study. The minimum sample size was calculated as 104 premature infants, with 26 infants per group, for a two-tailed hypothesis, an effect size of d = 0.929, an allocation ratio of 1:1, type I error of 0.05, and a power of 90%. Considering that there may be drop-outs during the process, the number of groups was increased by 20%. The sample size of this study was determined as 128 premature infants (32 premature infants in each intervention group).

Data Collection Tools Premature Infant's Information and Observation Form: This form was developed by the researchers after the literature review. It contains variables including gestational age at birth, postnatal age, birth weight, sex, procedural pain experience within the 24 hours prior to the intervention, the number of punctures performed during the intervention, duration of the intervention, duration of crying, the occurrence of adverse events during the intervention, heart rate, respiratory rate, saturation, and N-PASS score of premature infants before, during, and after the intervention.

Neonatal Pain Agitation and Sedation Scale - NPASS: Developed by Hummel et al. (2007, 2010), the Turkish validity-reliability study of this scale was conducted by Açıkgöz et al. (2017) and it is used for the quantitative assessment of acute, prolonged, chronic and postoperative pain in the first 100 days of life starting from the 23rd week of gestational age. The N-PASS is comprised of two measurements, each of which uses five criteria: crying/irritability, behavioral state, facial expression, extremity tone and vital signs. The pain score is assessed through observation without intervention, with a score range of 0 to 10, with 0 to 2 points available for each criterion. Points are added to the preterm infant's pain score (<28 weeks (3 points), 28-31 weeks (2 points), and 32-35 weeks (1 point)) to approximate the normal response of a full-term infant. Higher values represent higher pain.

Intervention: For each group, supportive positions are the facilitated flexion, nesting, and midline positions. Soft blankets and pillows will be used for positioning and nesting. The premature infants will be safely swaddled with a blanket supporting the natural fetal position that facilitated flexion and midline position. The enrolled premature infants will be administered 1ml of the oral solution a first time 2 minutes before the procedure. After 2 minutes, heel-stick sampling (with an auto lancet for premature infants) will be performed immediately after administering 1 ml of oral solution a second time. The infant's face and the monitor screen will be recorded in real-time using two independent video cameras during the entire procedure (starting 3 minutes prior to heel-stick sampling and continuing until the infant's crying is over). The N-PASS will be assessed during heel punction, at 1st minute, and 2nd minute after the procedure. After the end of the procedure, the recordings will be evaluated by two nurses, independent from each other. Oxygen saturation, heart rate and crying time will be determined from video recordings.

Ethical Considerations: The study was granted approval by the clinical research ethics committee and written institutional permission by the hospital. Parents will be informed about the procedure and written consent will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (GA) at birth 33+0 - 37+0 weeks
* Admitted to NICU
* Planned the heel-stick sampling within the scope of the NSTs
* Parents are able to read, write and speak Turkish

Exclusion Criteria:

* With a postnatal age of 8 days or more
* Has contraindications for the administration of oral glucose (genetic, endocrine, metabolic diseases or neurological problems etc.)
* Has major congenital anomalies
* Has intubated or receiving a nCPAP
* Has received analgesics or sedatives for less than 24 hours before the procedure

Ages: 2 Days to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Pain will be measured by N-PASS | at the heel punction during heel-stick sampling
  It is scored with 0 to 2 points available for each criterion (crying/irritability, behavioral state, facial expression, extremity tone and vital signs) and ranged from 0 to 10. Higher values represent higher pain.
Pain will be measured by N-PASS | at 1st minute after the heel punction
  It is scored with 0 to 2 points available for each criterion (crying/irritability, behavioral state, facial expression, extremity tone and vital signs) and ranged from 0 to 10. Higher values represent higher pain.
Pain will be measured by N-PASS | at 2st minute after the heel punction
  It is scored with 0 to 2 points available for each criterion (crying/irritability, behavioral state, facial expression, extremity tone and vital signs) and ranged from 0 to 10. Higher values represent higher pain.

SECONDARY OUTCOMES:
Duration of crying will be documented by video recordings | The total crying time is measured from where it starts until the over.
  Total amount of time (in minutes) the infant is crying during the procedure.

OTHER OUTCOMES:
Number of Participants with Adverse Events | Within 2 minutes following the procedure and oral solution
  Choking, coughing or vomiting Sustained tachycardia (HR>200) for >15 seconds Sustained bradycardia (HR<80) for >15 seconds Sustained tachypnea (RR>80) for >15 seconds Sustained dyspnea (RR<20) for >15 seconds Sustained oxygen desaturation <80% for >15 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Guzide UGUCU, Principal Investigator — Mersin University
Locations (1):
- Mersin University Hospital, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Result] Ugucu G, Yigit R, Celik Y. Effect of combining oral glucose solutions with supportive positions on pain during heel puncture blood sampling in premature infants: A randomized quadruple-blinded experimental study. J Pediatr Nurs. 2024 Jul-Aug;77:e108-e116. doi: 10.1016/j.pedn.2024.03.038. Epub 2024 Apr 3. PMID 38570229